CLINICAL TRIAL: NCT05336734
Title: Inter-Brain Synchrony in Psychotherapy for Test Anxiety
Acronym: IBSP-TA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 185/21
Record Dates: First submitted 2022-04-06; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Test Anxiety
Keywords: Synchrony; fNIRS; imaging; psychotherapy
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study was designed to examine changes in inter-brain synchrony over the course of standard psychotherapy, and not treatment effectiveness. As such, a single group design was deemed adequate.
Masking Description: There was no assignment to different groups and as a result, no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main group (Experimental): The group underwent a psychotherapy course combining CBT and imagery work. (For full protocol see Prinz et al., 2019)
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — see group description

SUMMARY:
The study aims to examine inter-brain synchrony between patients and therapists over the course of psychotherapy. Eight patients underwent a 6-session course of psychotherapy for test anxiety including Cognitive Behavioral Therapy (CBT) and imagery work, following an existing protocol (see Prinz et al., 2019), as well as a pre- and post- treatment interview (with different interviewers). The researchers used functional near-infrared spectroscopy (fNIRS) imaging to record brain activity during both interviews and sessions 1, 3, and 5, and collected saliva samples to measure hormone levels during the same sessions. Participants completed questionnaires before and after the study, and before and after each session.

The researchers hypothesized that synchrony will gradually increase over the psychotherapy sessions, that synchrony in the pre-treatment interview will be lower than in the post-treatment interview, and that synchrony would be correlated with increases in Oxytocin.

DETAILED DESCRIPTION:
This study centers on a short-term 6-session imagery-based treatment protocol for Test anxiety (Developed by Prof. Eshkol Rafaeli who is a collaborator on the study, with colleagues at the University of Trier; for the full protocol, see www.osf.io/hraqd). The protocol integrates traditional cognitive behavioral and imagery techniques; each session is also followed by some homework assignment, aimed at practicing the contents of the session and/or preparing for the next one.

The study lasted 8 weeks. On weeks 1 and 8 participants came in to a screening interview preformed by a research assistant. On weeks 2-7 participants came in to therapy meetings, according to the aforementioned protocol. On weeks 1,2,4,6,8 the researchers also performed functional near-infrared spectroscopy (fNIRS). imaging and took saliva samples. Participants, assessors (in assessment sessions) and therapists (in treatment sessions) underwent fNIRS imaging and provided saliva samples to measure Oxytocin and Cortisol levels. Samples were tested for hormonal levels and subsequently destroyed.

The study was an exploratory study, with the same therapist, who was a licensed clinical psychologist, treating all patients. He received supervision from an experienced psychologist with long experience employing cognitive-behavioral and experiential treatment methods.

Preliminary questionnaires. (a) Test Anxiety Inventory (b) Young Schema Questionnaire (YSQ-3) to assess early maladaptive schemas; (c) Ten Item Personality Inventory (TIPI) to assess Big-5 characteristics; (d) Schema Mode Inventory (SMI-2) to assess schema modes ; (e) Adult Attention Deficit Hyperactivity Disorder (ADHD) Self Report Scale; (f) Inventory of Interpersonal Problems (IIP) to assess interpersonal problems; (f) General Anxiety Disorder 7-item (GAD7) scale to assess anxiety symptoms; (g) Mindset questionnaire; (h) Patient Health Questionnaire (PHQ9) to assess depression symptoms; (i) Relationship Quality (RQ) to assess attachment; (j) demographic questionnaire; (k) Trauma questionnaires - The life event and Post Traumatic Stress Disorder checklists for the Diagnostic and Statistical Manual (DSM-5) and the Adverse Childhood Experiences Scale .

ELIGIBILITY:
Inclusion Criteria:

* Test Anxiety Inventory at least 50.

Exclusion Criteria:

* Participants with severe mood, anxiety, obsessional, psychotic, or eating disorders as assessed using a Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive and related Neuropsychiatric Disorders (DIAMOND) interview were excluded (However, comorbid single-episode major depressive disorder or social anxiety disorder did not lead to exclusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline State Test Anxiety | Weeks 2,7
  A six-item self-report questionnaire designed to measure test anxiety, evaluation apprehension and low efficacy (Lawrence & Williams, 2013). Change was defined as the difference between State Test Anxiety at week 7 and at week 2, and a successful outcome would be State Test Anxiety being lower at week 7 than at week 2. The scale is comprised of 6 items scored between 0 and 6, with the scale value being the mean of the items and as such also ranging between 0 and 6, with higher values representing more anxiety (i.e., more symptoms).

SECONDARY OUTCOMES:
Change from baseline Test Anxiety Inventory | Weeks 1,8
  A 20-item questionnaire measuring test anxiety (Spielberger, 1980). Change was defined as the difference between Test Anxiety Inventory values at week 1 and at week 8, and a successful outcome would be Test Anxiety Inventory being lower at week 8 than at week 1. Each item is scored between 1 and 4 and the scale value is calculated by summing the items, such that the scale ranges between 20 and 80, with high values representing more anxiety (i.e., more symptoms).

OTHER OUTCOMES:
Change from baseline Outcome Rating Scale | Weeks 2,7
  The Outcome Rating Scale (ORS) is a 4-item questionnaire evaluating general wellbeing (Miller et al., 2003). Change was defined as the difference between the ORS at week 7 and at week 2, and a successful outcome would be ORS at week 7 being higher than at week 2. ORS is presented as 4 visual slider items, and the scale is calculated by mapping each slider position to a number between 0 and 100 and calculating the mean of the 4 items, resulting in a scale ranging between 0 and 100 with 100 representing greater wellbeing.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Numerical questionnaire data, hormone levels and fNIRS recordings will be made available to other researchers.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication.
Access Criteria: Open Access

REFERENCES:
- [Background] Prinz JN, Bar-Kalifa E, Rafaeli E, Sened H, Lutz W. Imagery-based treatment for test anxiety: A multiple-baseline open trial. J Affect Disord. 2019 Feb 1;244:187-195. doi: 10.1016/j.jad.2018.10.091. Epub 2018 Oct 6. PMID 30343122
- [Background] Spielberger, C.D. Test anxiety inventory: Preliminary professional manual. Palo Alto,CA: Consulting Psychologist Press. 1980.
- [Background] Lawrence, J. S., & Williams, A. Anxiety explains why people with domain-contingent self-worth underperform on ability-diagnostic tests. Journal of Research in Personality. 2013; 47(3): 227-232